CLINICAL TRIAL: NCT05059535
Title: Cryoneurolysis of the Saphenous Nerve or Geniculate Nerves: Impact on Postoperative Pain and Rehabilitation in Prosthetic Knee Surgery
Brief Title: Knee Nerve Cryoneurolysis and Impact on Pain After Prosthetic Surgery
Acronym: Cryogenou
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: the recruitment rate is far too low despite an 18-month extension of the inclusion period
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-A01321-40
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cryoneurolysis of the saphenous nerve (Experimental): A cryoneurolysis of the saphenous nerve will be performed between 7 days and 5 days before the knee arthroplasty
  Interventions: Drug: standard pain relievers
- cryoneurolysis of geniculate nerves (Experimental): A cryoneurolysis of geniculate nerves will be performed between 7 days and 5 days before the knee arthroplasty
  Interventions: Drug: standard pain relievers
- control (Placebo Comparator): No cryoneurolysis will be performed before the knee arthroplasty
  Interventions: Drug: standard pain relievers

INTERVENTIONS:
Drug: standard pain relievers — Knee arthroscopy will be performed ansd patients will receive standard pain relievers in confomtity with the current practice
  Other Names: Standard pain relievers in accordance with the current practice

SUMMARY:
Interventional, comparative, randomized, controlled study versus standard treatment, in 3 parallel groups, monocentric, aiming to demonstrate the superiority of preoperative cryoneurolysis versus no procedure, in patients operated on for knee arthroplasty and receiving standard analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years;
* Patient to undergo prosthetic knee surgery;
* Patient in good health (ASA score 1 to 3);
* Patient able to understand the information related to the study, read the information leaflet and agree to sign the consent form.

Exclusion Criteria:

* Known intolerance to any of the products administered during surgery or cryoneurolysis;
* Patient with an electric implant;
* Patient with a contraindication to cryoanalgesia (coagulation disorders, infections, nerve damage);
* Drug addict patient;
* Intervention on septic bone;
* Chronic renal failure (creatinine clearance <30 mL / min);
* History of cryoglobulinemia, cold urticaria or Raynaud's syndrome;
* Pregnant or breastfeeding woman;
* Patient under guardianship or curatorship, or under a regime of deprivation of liberty;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient not beneficiary of a social security scheme.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
90 ° flexion pain 2 days after the arthroscopy | 2 days
  Evaluation of the knee pain at 90° flexion with a visual analogic scale of 100 mm

SECONDARY OUTCOMES:
90 ° flexion pain 1 day after the arthroscopy | 1 day
  Evaluation of the knee pain at 90° flexion with a visual analogic scale of 100 mm
90 ° flexion pain 7 days after the arthroscopy | 7 days
  Evaluation of the knee pain at 90° flexion with a visual analogic scale of 100 mm
90 ° flexion pain 30 days after the arthroscopy | 30 days
  Evaluation of the knee pain at 90° flexion with a visual analogic scale of 100 mm
90 ° flexion pain 90 days after the arthroscopy | 90 days
  Evaluation of the knee pain at 90° flexion with a visual analogic scale of 100 mm
pain at rest at Day 1 | 1 day
  Knee pain after intervention with a visual analogic scale of 100 mm
pain at rest at Day 2 | 2 days
  Knee pain after intervention with a visual analogic scale of 100 mm
pain at rest at Day 7 | 7 days
  Knee pain after intervention with a visual analogic scale of 100 mm
pain at rest at Day 30 | 30 days
  Knee pain after intervention with a visual analogic scale of 100 mm
pain at rest at Day 90 | 90 days
  Knee pain after intervention with a visual analogic scale of 100 mm

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé Paul d'Egine, Champigny-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No